CLINICAL TRIAL: NCT02007395
Title: Prospective Study on Polypectomy Complications: SPoC.
Status: Completed | Type: Observational
Sponsor: Valduce Hospital (Other)
Responsible Party: Principal Investigator, Arnaldo Amato, MD, Valduce Hospital
Other Study IDs: 5/2013
Record Dates: First submitted 2013-12-05; First posted 2013-12-10 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Endoscopic Polypectomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- colonoscopy population

SUMMARY:
Colonoscopy has been shown to reduce both the colo-rectal cancer incidence and mortality, due to its capability to detect and remove precancerous lesions. However, polypectomy is associated with complications, such as bleeding and perforation, with an estimated overall incidence of about 10%, with polyp size and right-sided location considered as major risk factors. Aim of present study was to prospectively evaluate the early and delayed (30-days follow-up) complications of polypectomy in a multicenter regional Italian real practice setting

ELIGIBILITY:
Inclusion Criteria:

* adult patients undergoing endoscopic polypectomy

Exclusion Criteria:

* pregnancy
* incapacity to give informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population undergoing endoscopic polypectomy
Sampling Method: Non-Probability Sample
Enrollment: 5170 (Actual)
Dates: Start 2013-06; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
complications of endoscopic polypectomy | 3 months